CLINICAL TRIAL: NCT07222683
Title: The Impact of Renal Transplant on Coronary Microvascular Function Among Patients With Advanced Chronic Kidney Disease
Acronym: RESTORE
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (AHA) (Unknown)
Responsible Party: Principal Investigator, Daniel Michael Huck, MD, MPH, Clinical Investigator, Brigham and Women's Hospital
Other Study IDs: 2022P002317; K23HL171893-01A1 (NIH)
Record Dates: First submitted 2025-10-27; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease; Kidney Transplant; Coronary Microvascular Dysfunction (CMD); Inflammation
Keywords: chronic kidney disease; coronary microvascular dysfunction; kidney transplant; cardiovascular inflammation; dysregulated angiogenesis; coronary artery disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (Plasma, Serum, Peripheral blood mononuclear cell PMBCs) and Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transplant Arm: Patients followed before and after transplant
- Waitlist Control Arm: Patients followed before transplant while on the waitlist

SUMMARY:
People with chronic kidney disease (CKD) often experience faster aging of the heart and blood vessels, which raises the risk of heart problems beyond traditional factors like high blood pressure or cholesterol. One early sign is reduced blood flow in the tiny vessels that supply the heart, measured by a positron emission tomography (PET) scan using a marker called myocardial flow reserve (MFR). In CKD, ongoing inflammation and abnormal blood vessel growth can damage these small vessels, leading to heart stiffness and weaker heart function.

A kidney transplant offers a unique chance to study how better kidney function and reduced inflammation affect heart health. The observational RESTORE study ("Impact of Renal Transplant on Coronary Microvascular Function in Patients with Advanced CKD") will measure heart blood flow and function before and after transplant.

The study will test whether:

1. Inflammation and abnormal vessel growth are linked to poor heart blood flow and heart function in CKD.
2. Kidney transplant improves heart blood flow and function.
3. Lower inflammation after transplant leads to better heart health.

By understanding how kidney disease and inflammation affect the heart-and how transplant may reverse these effects-this research could help guide future treatments to better protect heart health in patients with CKD.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant candidate on the waitlist
* Age greater or equal to 45 years, or if 18-44 years of age on dialysis for 5 years or more

Exclusion Criteria:

* Left ventricular ejection fraction (LVEF) < 40%
* History of coronary artery bypass grafting (CABG)
* History of heart transplant
* Patients who undergo revascularization as a result of pre-transplant cardiac PET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with advanced kidney disease who are candidates for renal transplant will be included in the RESTORE study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Stress Myocardial Blood Flow (MBF) | 1. Transplant Arm: At baseline prior to transplant and one year after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  Myocardial blood flow with hyperemic stress measured on PET myocardial perfusion imaging
Myocardial Flow Reserve (MFR) | 1. Transplant Arm: At baseline prior to transplant and one year after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  Ratio of stress and rest myocardial blood flow assessed by PET
Left ventricular global longitudinal strain (GLS, %) | 1. Transplant Arm: At baseline prior to transplant and one year after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  Left ventricular global longitudinal strain measured on echocardiography
Left ventricular mitral inflow velocity to mitral annular early diastolic relaxation velocity ration (E/E') | 1. Transplant Arm: At baseline prior to transplant and one year after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  E/E' measured by echocardiography
Interleukin-6 (IL-6) levels | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  IL-6 levels measured via proteomics assays
Vascular Endothelial Growth Factor A (VEGF-A) | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  VEGF-A measured by proteomic assay
Angiopoeitin-1 (ANGPT1) Levels | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  ANGPT1 levels measured by proteomic assay
Angiopoeitin-2 (ANGPT2) Levels | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  ANGPT2 levels measured by proteomics

SECONDARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | 1. Transplant Arm: At baseline prior to transplant and one year after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  LVEF by echocardiography
High sensitivity c-reactive protein (hs-CRP) | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  hs-CRP measured by blood assay
High-sensitivity Troponin | 1. Transplant Arm: At baseline prior to transplant, and 0, 2, 4, 6 and 12 months after transplant 2. Waitlist Control Arm: At baseline prior to transplant and one year after baseline while remaining on the transplant waitlist
  High-sensitivity troponin by blood assay

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All longitudinal human subjects data described in outcomes measures will be shared in a deidentified form. Both summarized data and individual will be shared via ClinicalTrials.gov and BioLINCC. Cardiovascular imaging data including PET and echocardiography will be shared as calculated parameters after expert interpretation from the raw images. The raw images will not be shared in a data depository, due to very large file-size, and the need for specialized software and expertise to interpret the imaging data. However, raw images may be available in a deidentified form upon appropriate and relevant request with an appropriate data transfer agreement. The protocol, sample informed consent, sample surveys, and data dictionaries will be shared on a data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Start Date: June 30, 2030 End Date: Indefinite ClinicalTrials.gov and BioLINCC will make decisions about how long to preserve the data, but no deposited data has been deleted up to now.
Access Criteria: All summarized and completely deidentified data on ClinicalTrials.gov will be publicly accessible without restriction. Data and metadata on the data repository BioLINCC will be controlled by standard processes at BioLINCC, including requirement for being a registered user on BioLINCC, the submission of an online request form, IRB approval, a research material distribution agreement, and approval by the NHLBI Data Repository Program Officer